CLINICAL TRIAL: NCT00576316
Title: Symbicort Maintenance And Reliever Therapy - Experience in Real Life Setting in Malaysia - SMARTER Study
Brief Title: Symbicort Maintenance and Reliever Therapy - Experience in Real Life Setting in Malaysia
Acronym: SMARTER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D5890L00027
Record Dates: First submitted 2007-12-17; First posted 2007-12-19 (Estimated); Results first posted 2009-12-29 (Estimated); Last update posted 2010-12-16 (Estimated); Status verified 2010-11

CONDITIONS: Asthma
Keywords: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Symbicort Turbuhaler 160/4.5

SUMMARY:
The purpose of the study is to evaluate the satisfaction level of patients using the Symbicort SMART approach for their asthma management.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of asthma for past 6 months and treated with inhaled glucocorticosteroids for at least 3 months.
* Patients who asthma is classified as uncontrolled or partially controlled as defined by GINA 2006 guidelines.

Exclusion Criteria:

* Patients already on Symbicort SMART treatment.
* Patients who has respiratory tract infection 30 days before study enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2008-01; Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Akhmal Yusof, MD, Study Director — AstraZeneca; Aziah Ahmad Mahayiddin, MD, Principal Investigator — Kuala Lumpur Hospital
Locations (1):
- Research Site, Kuala Lumpur, Malaysia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 201 patients were recruited from 10 government hospital based outpatient clinics from Dec 2007 until May 2008
Groups:
- Symbicort 160/4.5 Turbuhaler: Treatment with Symbicort 160/4.5 Turbuhaler 1 or 2 inhalations twice daily and when required as reliever
Period: Overall Study
Arm/Group | Symbicort 160/4.5 Turbuhaler
Started | 201 (Number of patients recruited)
Completed | 181 (Number of patients who completed study)
Not Completed | 20
Not completed — Adverse Event | 9
Not completed — Withdrawal by Subject | 2
Not completed — Protocol Violation | 9

BASELINE CHARACTERISTICS:
Arm/Group | Symbicort 160/4.5 Turbuhaler
Number analyzed (Participants) | 201
Age Continuous [Mean (Standard Deviation); unit: years]
  Mean Age | 46.73 (12.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 155
  Male | 46

OUTCOME MEASURES:

1. Primary Outcome: Change in Satisfaction With Asthma Treatment Questionnaire (SATQ) Scores From Baseline to the Mean of 3 Months and 6 Months After Patient Was Initially Treated With SMART
Description: Difference/change in SATQ score between baseline and mean of 3 months and 6 months after SMART treatment as analysed by paired t-test. SATQ is a patient reported questionnaire which consists of 26 questions and scored to a scale of 1-7, the higher score indicating a greater level of satisfaction
Time Frame: 6 months after each patient was initially treated with Symbicort SMART
Population: 201 participants were recruited but statistical analysis was completed for 195 participants
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Symbicort 160/4.5 Turbuhaler
Number analyzed (Participants) | 195
Scores on a scale | 0.37 (0.73)

2. Secondary Outcome: Changes in Asthma Control Questionnaire (ACQ-5) Score From Baseline to the Mean of 3 Months and 6 Months After Patient Was Initially Treated With SMART
Description: Difference/change in ACQ-5 scores between baseline and mean of 3 months and 6 months after SMART treatment. ACQ-5 is a 5 question patient reported outcome measuring level of asthma control during the past 7 days and it is scored on scale of 0-6. 0 indicates no symptoms and 6 represents severe symptoms
Time Frame: 6 months after each patient was initially treated with Symbicort SMART
Population: 201 participants were recruited but statistical analysis was completed for 195 participants
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Symbicort 160/4.5 Turbuhaler
Number analyzed (Participants) | 195
scores on a scale | -0.97 (1.22)

ADVERSE EVENTS:
Arm/Group | Symbicort 160/4.5 Turbuhaler
Serious Adverse Events (participants affected / at risk) | 17
Other Adverse Events (participants affected / at risk) | 70
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Symbicort 160/4.5 Turbuhaler
Congestive Cardiac Failure (Cardiac disorders) | 1/195
Vestibular Neuronitis (Ear and labyrinth disorders) | 1/195
Secretion And Pyrexia (General disorders) | 3/195
Upper Respiratory Tract Infection (Infections and infestations) | 5/195
Asthma (Respiratory, thoracic and mediastinal disorders) | 15/195
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Symbicort 160/4.5 Turbuhaler
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 26/195
General discomfort (General disorders) | 11/195
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 33/195

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less